CLINICAL TRIAL: NCT03022981
Title: A Phase 2, Open-Label, Multicenter, Multi-cohort Study to Investigate the Safety and Efficacy of Sofosbuvir/Velpatasvir in Adolescents and Children With Chronic HCV Infection
Brief Title: Study to Investigate the Safety and Efficacy of Sofosbuvir/Velpatasvir in Adolescents and Children With Chronic HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1143; 2016-002446-23 (EudraCT Number)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 12 to < 18 Years Old (Experimental): PK Lead-in Phase: Sofosbuvir/Velpatasvir (SOF/VEL) 400/100 mg once daily for 7 days. Participants who complete the PK lead-in phase, continue into the treatment phase with no interruption of study drug administration and additional participants will be enrolled into the treatment phase once the appropriateness of the dose is confirmed by PK results from the PK lead-in phase.
  Treatment Phase: SOF/VEL 400/100 mg once daily for 12 weeks.
  Interventions: Drug: SOF/VEL
- 6 to < 12 Years Old (Experimental): PK Lead-in Phase: SOF/VEL 200/50 mg once daily for 7 days. Participants who complete the PK lead-in phase, continue into the treatment phase with no interruption of study drug administration and additional participants will be enrolled into the treatment phase once the appropriateness of the dose is confirmed by PK results from the PK lead-in phase.
  Treatment Phase: SOF/VEL 200/50 mg once daily for 12 weeks.
  Interventions: Drug: SOF/VEL
- 3 to < 6 Years Old (Experimental): PK Lead-in Phase: SOF/VEL 200/50 mg once daily for 7 days for participants who weigh ≥ 17 kg. SOF/VEL 150/37.5 mg once daily for 7 days for participants who weigh < 17 kg. Participants who complete the PK lead-in phase, continue into the treatment phase with no interruption of study drug administration and additional participants will be enrolled into the treatment phase once the appropriateness of the dose is confirmed by PK results from the PK lead-in phase.
  Treatment Phase: SOF/VEL 200/50 mg once daily for 12 weeks for participants who weigh ≥ 17 kg. SOF/VEL 150/37.5 mg once daily for 12 weeks for participants who weigh < 17 kg.
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — SOF/VEL fixed-dose combination (FDC) 400/100 mg tablets or SOF/VEL FDC 200/50 mg tablets (based on swallowability assessment)
  Other Names: Epclusa®; GS-7977/GS-5816
  Arms: 12 to < 18 Years Old; 6 to < 12 Years Old
Drug: SOF/VEL — SOF/VEL FDC 200/50 mg oral granules
  Other Names: Epclusa®; GS-7977/GS-5816
  Arms: 3 to < 6 Years Old

SUMMARY:
This study will have 2 parts: Pharmacokinetics (PK) Lead-in Phase and the Treatment Phase.

The primary objective of the PK Lead-in Phase is to evaluate the steady state PK and confirm the dose of sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) in pediatric participants with chronic hepatitis C virus (HCV) infection.

The primary objective of the Treatment Phase is to evaluate the safety and tolerability of SOF/VEL for 12 weeks in pediatric participants with chronic HCV.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic HCV-infected, treatment-naive and treatment-experienced adolescent and pediatric individuals aged 3 to < 18 as determined at Day 1.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (27):
- United States (21):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Medical, Gainesville, Florida
  - Florida Gastroenterology Care for Children, Orlando, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Johns Hopkins University (JHU) - The Johns Hopkins Hospital (JHH), Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital- The Ohio State University (OSU), Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Cliniques Universitaires Saint Luc, Brussels, Belgium
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Meyer, Florence
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- United Kingdom (2):
  - The Leeds Teaching Hospitals NHS Trust, Leeds, England
  - King's College Hospital NHS Trust, London, England

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Jonas MM, Romero R, Sokal EM, Rosenthal P, Verucchi G, Lin CH, et al. The Safety and Efficacy of Sofosbuvir/Velpatasvir in Pediatric Patients 6 to < 18 years old with Chronic Hepatitis C Infection [Abstract]. AASLD; 2019 08-12 November; Boston, Massachusetts.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 28 study sites in Belgium, Italy, the United Kingdom, and the United States. The first participant was screened on 26 January 2017. The last study visit occurred on 26 February 2020.
Pre-assignment Details: 221 participants were screened.
Groups:
- 12 to < 18 Years Old: Pharmacokinetic (PK) Lead-in Phase: Sofosbuvir/Velpatasvir (SOF/VEL) fixed-dose combination (FDC) 400/100 mg tablets once daily for 7 days. Participants who completed the PK lead-in phase, continued into the treatment phase with no interruption of study drug administration and additional participants were enrolled into the treatment phase once the appropriateness of the dose was confirmed by PK results from the PK lead-in phase.
  Treatment Phase: SOF/VEL 400/100 mg (adult and smaller size tablets based on swallowability assessment) once daily for 12 weeks.
- 6 to < 12 Years Old: PK Lead-in Phase: SOF/VEL FDC 200/50 mg tablets or oral granules once daily for 7 days. Participants who completed the PK lead-in phase, continued into the treatment phase with no interruption of study drug administration and additional participants were enrolled into the treatment phase once the appropriateness of the dose was confirmed by PK results from the PK lead-in phase.
  Treatment Phase: SOF/VEL FDC 200/50 mg tablets or oral granules once daily for 12 weeks.
- 3 to < 6 Years Old: PK Lead-in Phase: SOF/VEL FDC 200/50 mg oral granules once daily for 7 days for participants who weighed ≥ 17 kg. SOF/VEL FDC 150/37.5 mg oral granules once daily for 7 days for participants who weighed < 17 kg. Participants who completed the PK lead-in phase, continued into the treatment phase with no interruption of study drug administration and additional participants were enrolled into the treatment phase once the appropriateness of the dose was confirmed by PK results from the PK lead-in phase.
  Treatment Phase: SOF/VEL FDC 200/50 mg oral granules once daily for 12 weeks for participants who weighed ≥ 17 kg. SOF/VEL FDC 150/37.5 mg oral granules once daily for 12 weeks for participants who weighed < 17 kg.
Period: Overall Study
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Started | 102 | 73 | 41
Participated in PK Lead-in (PKL) Phase | 17 (All 17 participants completed treatment in the PK Lead-in phase and continued into treatment phase.) | 20 (All 20 participants completed treatment in the PK Lead-in phase and continued into treatment phase.) | 19 (All 19 participants completed treatment in the PK Lead-in phase and continued into treatment phase.)
Completed | 96 | 69 | 35
Not Completed | 6 | 4 | 6
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Investigator's Discretion | 0 | 1 | 2
Not completed — Lost to Follow-up | 6 | 2 | 1
Not completed — Non-Compliance With Study Drug | 0 | 0 | 2
Not completed — Withdrew Assent By Parent/Guardian | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug (SOF/VEL FDC).
Groups:
- 12 to < 18 Years Old: PK Lead-in Phase: Sofosbuvir/Velpatasvir (SOF/VEL) fixed-dose combination (FDC) 400/100 mg tablets once daily for 7 days. Participants who completed the PK lead-in phase, continued into the treatment phase with no interruption of study drug administration and additional participants were enrolled into the treatment phase once the appropriateness of the dose was confirmed by PK results from the PK lead-in phase.
  Treatment Phase: SOF/VEL 400/100 mg (adult and smaller size tablets based on swallowability assessment) once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old | Total
Number analyzed (Participants) | 102 | 73 | 41 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.9) | 8 (1.6) | 4 (0.8) | 10 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 38 | 24 | 114
  Male | 50 | 35 | 17 | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local requirements did not permit collection of race or ethnicity information.
  Participants
    Race: White | 74 | 66 | 32 | 172
    Race: Black or African American | 9 | 4 | 3 | 16
    Race: Asian | 11 | 1 | 0 | 12
    Race: Other | 5 | 2 | 5 | 12
    Race: American Indian or Alaska Native | 2 | 0 | 0 | 2
    Race: Not Permitted | 1 | 0 | 1 | 2
    Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local requirements did not permit collection of race or ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 14 | 7 | 4 | 25
    Ethnicity: Not Hispanic or Latino | 83 | 64 | 36 | 183
    Ethnicity: Not Permitted | 5 | 2 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77 | 57 | 38 | 172
  Italy | 17 | 5 | 2 | 24
  United Kingdom | 5 | 9 | 1 | 15
  Belgium | 3 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: PK Lead-in Phase: AUCtau: Area Under the Plasma Concentration Versus Time Curve Over the Dosing Interval of Velpatasvir (VEL)
Description: AUCtau is defined as concentration of drug over time (the area under the concentration versus time curve over the dosing interval).
Time Frame: Day 7: 0 (predose), 0.5, 1, 2, 3, 4, 6 (Cohorts 1 and 2 only), 8, and 12 hours postdose
Population: The Lead-in Phase Pharmacokinetic (PK) Analysis Set included all PK lead-in phase participants with available data who received at least 1 dose of study drug and whom at least one non-missing PK concentration data value is available from the PK Lead-in Phase intensive sampling.
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter (h*ng/mL)
Groups:
- 12 to < 18 Years Old: PK Lead-in Phase: Sofosbuvir/Velpatasvir (SOF/VEL) fixed-dose combination (FDC) 400/100 mg tablets once daily for 7 days.
- 6 to < 12 Years Old: PK Lead-in Phase: SOF/VEL FDC 200/50 mg tablets or oral granules once daily for 7 days.
- 3 to < 6 Years Old: PK Lead-in Phase: SOF/VEL FDC 200/50 mg oral granules once daily for 7 days for participants who weighed ≥ 17 kg. SOF/VEL FDC 150/37.5 mg oral granules once daily for 7 days for participants who weighed < 17 kg.
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 16 | 17 | 18
hours*nanograms per milliliter (h*ng/mL) | 4479.3 (2105.66) | 3697.5 (1653.25) | 4450.3 (3285.75)

2. Primary Outcome: PK Lead-in Phase: AUCtau: Area Under the Plasma Concentration Versus Time Curve Over the Dosing Interval of Sofosbuvir (SOF)
Description: as for outcome 1
Time Frame: Day 7: 0 (predose), 0.5, 1, 2, 3, 4, 6 (Cohorts 1 and 2 only), 8, and 12 hours postdose
Population: Participants in the Lead-in Phase PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 12 to < 18 Years Old: PK Lead-in Phase: SOF/VEL FDC 400/100 mg tablets once daily for 7 days.
- Cohort 3 (3 to < 6 Years Old): PK Lead-in Phase: SOF/VEL FDC 200/50 mg oral granules once daily for 7 days for participants who weighed ≥ 17 kg. SOF/VEL FDC 150/37.5 mg oral granules once daily for 7 days for participants who weighed < 17 kg.
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | Cohort 3 (3 to < 6 Years Old)
Number analyzed (Participants) | 16 | 17 | 17
h*ng/mL | 3020.1 (1162.56) | 1764.5 (690.12) | 3306.2 (3499.49)

3. Primary Outcome: PK Lead-in Phase: AUCtau: Area Under the Plasma Concentration Versus Time Curve Over the Dosing Interval of GS-331007 (Metabolite of SOF)
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Day 7: 0 (predose), 0.5, 1, 2, 3, 4, 6 (Cohorts 1 and 2 only), 8, and 12 hours postdose
Population: Participants in the Lead-in Phase PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 16 | 17 | 18
h*ng/mL | 13852.9 (3565.85) | 9913.8 (3071.79) | 11604.0 (2732.57)

4. Primary Outcome: Treatment Phase: Percentage of Participants Who Discontinued Study Drug Due to Any Treatment-Emergent Adverse Event (TEAE)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs were defined as 1 or both of the following: Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and/or Any AEs leading to premature discontinuation of study drug.
Time Frame: From first dose through last dose of the study drug (Up to 12 weeks) plus 30 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- 12 to < 18 Years Old: Treatment Phase: SOF/VEL 400/100 mg (adult and smaller size tablets based on swallowability assessment) once daily for 12 weeks.
- 6 to < 12 Years Old: Treatment Phase: SOF/VEL FDC 200/50 mg tablets or oral granules once daily for 12 weeks.
- 3 to < 6 Years Old: Treatment Phase: SOF/VEL FDC 200/50 mg oral granules once daily for 12 weeks for participants who weighed ≥ 17 kg. SOF/VEL FDC 150/37.5 mg oral granules once daily for 12 weeks for participants who weighed < 17 kg.
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
percentage of participants | 0.0 | 2.7 | 2.4

5. Secondary Outcome: PK Lead-in Phase: Change From Baseline in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Day 7
Time Frame: Baseline; Day 7
Population: Participants in the Lead-in Phase PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 international units per mL (IU/mL)
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 17 | 20 | 19
log10 international units per mL (IU/mL)
  Baseline | 6.09 (0.569) | 5.84 (0.656) | 5.77 (1.275)
  Change from Baseline at Day 7 | -4.48 (0.656) | -4.20 (0.642) | -3.94 (1.082)

6. Secondary Outcome: PK Lead-in Phase: Percentage of Participants Who Permanently Discontinued Study Drug Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: First dose date up to Day 7
Population: Participants in the Lead-in Phase PK Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 17 | 20 | 19
percentage of participants | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Treatment Phase: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: The Full Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug (SOF/VEL FDC).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
percentage of participants | 95.1 [88.9 to 98.4] | 93.2 [84.7 to 97.7] | 82.9 [67.9 to 92.8]

8. Secondary Outcome: Treatment Phase: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ (ie, 15 IU/mL) at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
percentage of participants | 96.1 [90.3 to 98.9] | 94.5 [86.6 to 98.5] | 82.9 [67.9 to 92.8]

9. Secondary Outcome: Treatment Phase: Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR 24 was defined as HCV RNA < LLOQ (ie, 15 IU/mL) at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
percentage of participants | 95.1 [88.9 to 98.4] | 93.2 [84.7 to 97.7] | 82.9 [67.9 to 92.8]

10. Secondary Outcome: Treatment Phase: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as: On-treatment virologic failure - Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment); Virologic relapse: Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
percentage of participants | 1.0 | 1.4 | 0.0

11. Secondary Outcome: Treatment Phase: Percentage of Participants With HCV RNA < LLOQ On Treatment
Description: Percentage of participants with HCV RNA < LLOQ while on treatment by analysis visit.
Time Frame: Weeks 1, 4, 8, and 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
percentage of participants
  Week 1 | 44.1 [34.3 to 54.3] | 39.7 [28.5 to 51.9] | 36.8 [21.8 to 54.0]
  Week 4 | 96.1 [90.3 to 98.9] | 94.4 [86.2 to 98.4] | 91.4 [76.9 to 98.2]
  Week 8 | 100.0 [96.4 to 100.0] | 98.6 [92.3 to 100.0] | 100.0 [89.7 to 100.0]
  Week 12 | 100.0 [96.4 to 100.0] | 98.6 [92.3 to 100.0] | 100.0 [89.7 to 100.0]

12. Secondary Outcome: Treatment Phase: Percentage of Participants Who Develop Viral Resistance to SOF and/or VEL During Treatment and After Discontinuation of Treatment
Description: Drug-resistant substitutions were analyzed as part of the Virology Study. Plasma samples were collected and stored for potential HCV sequencing. Impact on the treatment outcomes of SVR12 and SVR24 were observed during the study. Baseline deep sequencing of the HCV nonstructural protein (NS)5A and NS5B genes was performed for all participants at the first time point after virologic failure if the plasma or serum sample was available. Pretreatment full-length NS5A deep sequencing data were obtained at a 15% assay cutoff for the Resistance Analysis Population which covered all NS5A and NS5B nucleoside inhibitor (NI) resistance-associated variants (RAVs).
Time Frame: First dose date up to Posttreatment Week 24
Population: The Resistance Analysis Population with all adolescent or pediatric participants in the Safety Analysis Set with a virologic outcome with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 98 | 68 | 33
percentage of participants
  Pretreatment NS5A NI RAVs | 16.3 | 10.2 | 18.1
  Pretreatment NS5B NI RAVs: number analyzed (Participants) | 66 | 68 | 33
  Pretreatment NS5B NI RAVs | 5.1 | 0.0 | 3.0

13. Secondary Outcome: Treatment Phase: Change From Baseline in HCV RNA at Weeks 1, 4, 8, and 12
Time Frame: Baseline; Weeks 1, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
log10 IU/mL
  Baseline | 6.06 (0.585) | 5.87 (0.686) | 5.86 (1.057)
  Change from Baseline at Week 1: number analyzed (Participants) | 102 | 71 | 36
  Change from Baseline at Week 1 | -4.46 (0.661) | -4.28 (0.632) | -4.06 (0.914)
  Change from Baseline at Week 4: number analyzed (Participants) | 102 | 71 | 34
  Change from Baseline at Week 4 | -4.89 (0.578) | -4.64 (0.860) | -4.49 (1.040)
  Change from Baseline at Week 8: number analyzed (Participants) | 101 | 70 | 34
  Change from Baseline at Week 8 | -4.91 (0.588) | -4.69 (0.678) | -4.56 (1.066)
  Change from Baseline at Week 12: number analyzed (Participants) | 101 | 69 | 34
  Change from Baseline at Week 12 | -4.91 (0.588) | -4.70 (0.683) | -4.56 (1.066)

14. Secondary Outcome: Treatment Phase: Quality of Life (QoL) and Neuropsychiatric Assessments as Measured by PedsQL™ Pediatric QoL Survey
Description: To evaluate the effect of treatment with SOF/VEL on general and disease-specific health-related QoL, the PedsQL™ Pediatric QoL Inventory V4.0 Short Form (SF15) was completed at Day 1, end of treatment, early termination (if applicable), and posttreatment Weeks 12 and 24. The SF15 questionnaire represented 4 domains: physical, emotional, social, and school functioning, with the emotional, social, and school functioning domains representing the psychosocial health summary. Neuropsychiatric assessment was conducted using the PedsQL™ Pediatric QoL Inventory V4.0 SF15 psychosocial domain-related scores. Items were calculated and transformed into an overall score with a range of 0 to 100 points, with more points indicating better QoL.
Time Frame: Baseline; Week 12, End of Treatment (EOT), Posttreatment/Follow-up (FU) Week-12 (FU-12), and FU Week-24 (FU-24)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
score on a scale
  Parents Reports, Total Score at Baseline: number analyzed (Participants) | 98 | 73 | 41
  Parents Reports, Total Score at Baseline | 80.0 (17.71) | 79.7 (15.58) | 86.5 (12.43)
  Parents Reports, Total Score at Week 12: number analyzed (Participants) | 97 | 68 | 32
  Parents Reports, Total Score at Week 12 | 82.4 (18.13) | 82.8 (14.26) | 87.3 (11.31)
  Parents Reports, Total Score at EOT: number analyzed (Participants) | 97 | 70 | 34
  Parents Reports, Total Score at EOT | 82.4 (18.13) | 82.2 (14.95) | 87.0 (11.65)
  Parents Reports, Total Score at Follow Up-12: number analyzed (Participants) | 94 | 68 | 35
  Parents Reports, Total Score at Follow Up-12 | 81.7 (17.39) | 81.5 (15.34) | 87.7 (14.11)
  Parents Reports, Total Score at Follow Up-24: number analyzed (Participants) | 94 | 69 | 35
  Parents Reports, Total Score at Follow Up-24 | 80.8 (18.65) | 79.7 (15.30) | 88.3 (9.79)
  Participants Reports, Total Score at Baseline: number analyzed (Participants) | 100 | 73 | 18
  Participants Reports, Total Score at Baseline | 79.9 (15.22) | 77.9 (13.33) | 82.2 (12.47)
  Participants Reports, Total Score at Week 12: number analyzed (Participants) | 101 | 68 | 21
  Participants Reports, Total Score at Week 12 | 80.9 (16.38) | 80.0 (14.21) | 83.3 (11.62)
  Participants Reports, Total Score at EOT: number analyzed (Participants) | 101 | 70 | 21
  Participants Reports, Total Score at EOT | 80.9 (16.38) | 79.7 (14.13) | 83.3 (11.62)
  Participants Reports, Total Score at Follow Up-12: number analyzed (Participants) | 98 | 68 | 23
  Participants Reports, Total Score at Follow Up-12 | 82.5 (15.41) | 81.1 (13.32) | 80.5 (14.18)
  Participants Reports, Total Score at Follow Up-24: number analyzed (Participants) | 98 | 69 | 25
  Participants Reports, Total Score at Follow Up-24 | 81.4 (16.34) | 81.7 (15.43) | 82.1 (12.56)

15. Secondary Outcome: Treatment Phase: Change From Baseline in Growth and Development as Measured by Height Percentiles
Description: An age- and sex-specific percentile was derived for each weight, height, and body mass index (BMI) measurement according to the statistical analysis system (SAS) program available on the Centers for Disease Control and Prevention (CDC) website using the year 2000 growth charts.
Time Frame: Baseline; Weeks 1, 4, 8, 12, Follow-up (FU) Week 4 (FU-4), FU-12, and FU-24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentile
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
percentile
  Baseline | 44.5 [16.2 to 74.1] | 41.9 [20.5 to 65.2] | 39.3 [13.9 to 70.1]
  Change From Baseline at Week 1: number analyzed (Participants) | 102 | 73 | 36
  Change From Baseline at Week 1 | 0.0 [-0.4 to 0.9] | 0.1 [-0.7 to 2.4] | 0.5 [-1.1 to 3.4]
  Change From Baseline at Week 4: number analyzed (Participants) | 101 | 71 | 34
  Change From Baseline at Week 4 | 0.0 [-0.7 to 1.7] | 0.2 [-1.9 to 1.9] | 1.4 [-0.3 to 3.7]
  Change From Baseline at Week 8: number analyzed (Participants) | 101 | 69 | 34
  Change From Baseline at Week 8 | 0.0 [-1.2 to 1.5] | -0.1 [-2.2 to 2.2] | 0.3 [-2.1 to 3.6]
  Change From Baseline at Week 12: number analyzed (Participants) | 100 | 65 | 28
  Change From Baseline at Week 12 | -0.1 [-1.4 to 1.0] | 0.2 [-2.6 to 2.8] | 0.2 [-2.0 to 5.1]
  Change From Baseline at FU-4: number analyzed (Participants) | 99 | 70 | 34
  Change From Baseline at FU-4 | 0.0 [-2.0 to 1.3] | 0.2 [-2.3 to 2.5] | 1.2 [-0.7 to 5.6]
  Change From Baseline at FU-12: number analyzed (Participants) | 98 | 68 | 35
  Change From Baseline at FU-12 | -0.2 [-2.4 to 1.4] | 0.1 [-1.7 to 2.6] | 0.6 [-3.1 to 4.6]
  Change From Baseline at FU-24: number analyzed (Participants) | 91 | 67 | 33
  Change From Baseline at FU-24 | -0.6 [-2.6 to 1.9] | -0.2 [-3.1 to 3.5] | 0.3 [-2.1 to 6.0]

16. Secondary Outcome: Treatment Phase: Change From Baseline in Growth and Development as Measured by Weight Percentiles
Description: An age- and sex-specific percentile was derived for each weight, height, and BMI measurement according to the SAS program available on the CDC website using the year 2000 growth charts.
Time Frame: Baseline; Weeks 1, 4, 8, 12, FU-4, FU-12, and FU-24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentile
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
percentile
  Baseline | 67.2 [31.5 to 84.1] | 45.9 [23.3 to 78.6] | 64.6 [38.0 to 86.7]
  Change From Baseline at Week 1: number analyzed (Participants) | 102 | 73 | 36
  Change From Baseline at Week 1 | 0.0 [-0.4 to 0.9] | 0.1 [-0.6 to 1.2] | -0.5 [-2.7 to 0.7]
  Change From Baseline at Week 4: number analyzed (Participants) | 102 | 71 | 34
  Change From Baseline at Week 4 | 0.0 [-0.9 to 1.8] | 0.2 [-1.4 to 1.5] | 0.3 [-1.2 to 2.0]
  Change From Baseline at Week 8: number analyzed (Participants) | 101 | 69 | 34
  Change From Baseline at Week 8 | 0.0 [-1.3 to 2.1] | 0.1 [-1.6 to 2.5] | 0.2 [-3.7 to 2.5]
  Change From Baseline at Week 12: number analyzed (Participants) | 100 | 65 | 28
  Change From Baseline at Week 12 | 0.2 [-1.0 to 2.9] | 0.5 [-1.7 to 2.5] | -1.7 [-4.7 to 0.6]
  Change From Baseline at FU-4: number analyzed (Participants) | 99 | 70 | 34
  Change From Baseline at FU-4 | 0.1 [-3.0 to 3.1] | 0.0 [-2.3 to 2.6] | -0.8 [-4.9 to 2.4]
  Change From Baseline at FU-12: number analyzed (Participants) | 98 | 68 | 35
  Change From Baseline at FU-12 | 0.0 [-2.5 to 4.7] | 0.5 [-2.2 to 4.9] | -0.8 [-6.6 to 2.2]
  Change From Baseline at FU-24: number analyzed (Participants) | 91 | 67 | 33
  Change From Baseline at FU-24 | 0.1 [-2.6 to 4.1] | 1.4 [-1.2 to 5.7] | -1.3 [-3.5 to 2.9]

17. Secondary Outcome: Treatment Phase: Changes in Growth and Development as Measured by Tanner Stage Assessment From Baseline
Description: Tanner Pubertal Staging was assessed for pubic hair growth and genitalia development (males) and for pubic hair growth and breast development (females) in stages 1 to 5. Tanner stages were used to evaluate the onset and progression of pubertal changes from stage 1 (pre-pubertal) to stage 5 (adult). If a participant had reached Tanner stage 5, no further Tanner pubertal stage assessments were to be completed. Pubic hair growth: Tanner stages (1: No hair, 2: Downy hair, 3: More coarse and curly hair, 4: Adult-like hair quality; 5: Hair extends to the medial surface of the thighs); Breast development: Tanner stages (1: No glandular tissue, 2: Breast bud forms,3: More elevated, outside areola, 4: Increased breast size,5: Final adult-size breasts); Genitalia development: Tanner stages (1: Testes, scrotum, and penis about same size, 2: Enlargement of scrotum, testes and penis, 3: Enlargement of penis, 4: Penis size enlargement, 5: Genitalia adult in size and shape).
Time Frame: Baseline; EOT, FU-12 and FU-24
Population: Participants in the Safety Analysis Set with available data were analyzed. Overall Number of Participants Analyzed for each arm is the total of male plus female participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
Participants
  Pubic Hair (Male): Baseline, Stage 1: number analyzed (Participants) | 50 | 34 | 17
  Pubic Hair (Male): Baseline, Stage 1 | 4 | 31 | 17
  Pubic Hair (Male): Baseline, Stage 2: number analyzed (Participants) | 50 | 34 | 17
  Pubic Hair (Male): Baseline, Stage 2 | 3 | 2 | 0
  Pubic Hair (Male): Baseline, Stage 3: number analyzed (Participants) | 50 | 34 | 17
  Pubic Hair (Male): Baseline, Stage 3 | 10 | 1 | 0
  Pubic Hair (Male): Baseline, Stage 4: number analyzed (Participants) | 50 | 34 | 17
  Pubic Hair (Male): Baseline, Stage 4 | 14 | 0 | 0
  Pubic Hair (Male): Baseline, Stage 5: number analyzed (Participants) | 50 | 34 | 17
  Pubic Hair (Male): Baseline, Stage 5 | 19 | 0 | 0
  Pubic Hair (Male): EOT, Stage 1: number analyzed (Participants) | 50 | 32 | 13
  Pubic Hair (Male): EOT, Stage 1 | 2 | 28 | 13
  Pubic Hair (Male): EOT, Stage 2: number analyzed (Participants) | 50 | 32 | 13
  Pubic Hair (Male): EOT, Stage 2 | 4 | 3 | 0
  Pubic Hair (Male): EOT, Stage 3: number analyzed (Participants) | 50 | 32 | 13
  Pubic Hair (Male): EOT, Stage 3 | 7 | 1 | 0
  Pubic Hair (Male): EOT, Stage 4: number analyzed (Participants) | 50 | 32 | 13
  Pubic Hair (Male): EOT, Stage 4 | 13 | 0 | 0
  Pubic Hair (Male): EOT, Stage 5: number analyzed (Participants) | 50 | 32 | 13
  Pubic Hair (Male): EOT, Stage 5 | 24 | 0 | 0
  Pubic Hair (Male): FU-12, Stage 1: number analyzed (Participants) | 47 | 30 | 14
  Pubic Hair (Male): FU-12, Stage 1 | 1 | 26 | 14
  Pubic Hair (Male): FU-12, Stage 2: number analyzed (Participants) | 47 | 30 | 14
  Pubic Hair (Male): FU-12, Stage 2 | 5 | 3 | 0
  Pubic Hair (Male): FU-12, Stage 3: number analyzed (Participants) | 47 | 30 | 14
  Pubic Hair (Male): FU-12, Stage 3 | 6 | 1 | 0
  Pubic Hair (Male): FU-12, Stage 4: number analyzed (Participants) | 47 | 30 | 14
  Pubic Hair (Male): FU-12, Stage 4 | 10 | 0 | 0
  Pubic Hair (Male): FU-12, Stage 5: number analyzed (Participants) | 47 | 30 | 14
  Pubic Hair (Male): FU-12, Stage 5 | 25 | 0 | 0
  Pubic Hair (Male): FU-24, Stage 1: number analyzed (Participants) | 45 | 32 | 14
  Pubic Hair (Male): FU-24, Stage 1 | 1 | 29 | 14
  Pubic Hair (Male): FU-24, Stage 2: number analyzed (Participants) | 45 | 32 | 14
  Pubic Hair (Male): FU-24, Stage 2 | 4 | 2 | 0
  Pubic Hair (Male): FU-24, Stage 3: number analyzed (Participants) | 45 | 32 | 14
  Pubic Hair (Male): FU-24, Stage 3 | 2 | 1 | 0
  Pubic Hair (Male): FU-24, Stage 4: number analyzed (Participants) | 45 | 32 | 14
  Pubic Hair (Male): FU-24, Stage 4 | 13 | 0 | 0
  Pubic Hair (Male): FU-24, Stage 5: number analyzed (Participants) | 45 | 32 | 14
  Pubic Hair (Male): FU-24, Stage 5 | 25 | 0 | 0
  Genitalia (Male): Baseline, Stage 1: number analyzed (Participants) | 50 | 34 | 17
  Genitalia (Male): Baseline, Stage 1 | 4 | 31 | 17
  Genitalia (Male): Baseline, Stage 2: number analyzed (Participants) | 50 | 34 | 17
  Genitalia (Male): Baseline, Stage 2 | 3 | 2 | 0
  Genitalia (Male): Baseline, Stage 3: number analyzed (Participants) | 50 | 34 | 17
  Genitalia (Male): Baseline, Stage 3 | 8 | 1 | 0
  Genitalia (Male): Baseline, Stage 4: number analyzed (Participants) | 50 | 34 | 17
  Genitalia (Male): Baseline, Stage 4 | 16 | 0 | 0
  Genitalia (Male): Baseline, Stage 5: number analyzed (Participants) | 50 | 34 | 17
  Genitalia (Male): Baseline, Stage 5 | 19 | 0 | 0
  Genitalia (Male): EOT, Stage 1: number analyzed (Participants) | 50 | 32 | 13
  Genitalia (Male): EOT, Stage 1 | 2 | 28 | 13
  Genitalia (Male): EOT, Stage 2: number analyzed (Participants) | 50 | 32 | 13
  Genitalia (Male): EOT, Stage 2 | 3 | 3 | 0
  Genitalia (Male): EOT, Stage 3: number analyzed (Participants) | 50 | 32 | 13
  Genitalia (Male): EOT, Stage 3 | 7 | 1 | 0
  Genitalia (Male): EOT, Stage 4: number analyzed (Participants) | 50 | 32 | 13
  Genitalia (Male): EOT, Stage 4 | 15 | 0 | 0
  Genitalia (Male): EOT, Stage 5: number analyzed (Participants) | 50 | 32 | 13
  Genitalia (Male): EOT, Stage 5 | 23 | 0 | 0
  Genitalia (Male): FU-12, Stage 1: number analyzed (Participants) | 47 | 30 | 14
  Genitalia (Male): FU-12, Stage 1 | 1 | 26 | 14
  Genitalia (Male): FU-12, Stage 2: number analyzed (Participants) | 47 | 30 | 14
  Genitalia (Male): FU-12, Stage 2 | 4 | 3 | 0
  Genitalia (Male): FU-12, Stage 3: number analyzed (Participants) | 47 | 30 | 14
  Genitalia (Male): FU-12, Stage 3 | 7 | 1 | 0
  Genitalia (Male): FU-12, Stage 4: number analyzed (Participants) | 47 | 30 | 14
  Genitalia (Male): FU-12, Stage 4 | 11 | 0 | 0
  Genitalia (Male): FU-12, Stage 5: number analyzed (Participants) | 47 | 30 | 14
  Genitalia (Male): FU-12, Stage 5 | 24 | 0 | 0
  Genitalia (Male): FU-24, Stage 1: number analyzed (Participants) | 45 | 32 | 14
  Genitalia (Male): FU-24, Stage 1 | 1 | 27 | 14
  Genitalia (Male): FU-24, Stage 2: number analyzed (Participants) | 45 | 32 | 14
  Genitalia (Male): FU-24, Stage 2 | 2 | 4 | 0
  Genitalia (Male): FU-24, Stage 3: number analyzed (Participants) | 45 | 32 | 14
  Genitalia (Male): FU-24, Stage 3 | 4 | 1 | 0
  Genitalia (Male): FU-24, Stage 4: number analyzed (Participants) | 45 | 32 | 14
  Genitalia (Male): FU-24, Stage 4 | 13 | 0 | 0
  Genitalia (Male): FU-24, Stage 5: number analyzed (Participants) | 45 | 32 | 14
  Genitalia (Male): FU-24, Stage 5 | 25 | 0 | 0
  Pubic Hair (Female): Baseline, Stage 1: number analyzed (Participants) | 52 | 38 | 24
  Pubic Hair (Female): Baseline, Stage 1 | 2 | 31 | 24
  Pubic Hair (Female): Baseline, Stage 2: number analyzed (Participants) | 52 | 38 | 24
  Pubic Hair (Female): Baseline, Stage 2 | 3 | 5 | 0
  Pubic Hair (Female): Baseline, Stage 3: number analyzed (Participants) | 52 | 38 | 24
  Pubic Hair (Female): Baseline, Stage 3 | 9 | 2 | 0
  Pubic Hair (Female): Baseline, Stage 4: number analyzed (Participants) | 52 | 38 | 24
  Pubic Hair (Female): Baseline, Stage 4 | 16 | 0 | 0
  Pubic Hair (Female): Baseline, Stage 5: number analyzed (Participants) | 52 | 38 | 24
  Pubic Hair (Female): Baseline, Stage 5 | 22 | 0 | 0
  Pubic Hair (Female): EOT, Stage 1: number analyzed (Participants) | 50 | 37 | 21
  Pubic Hair (Female): EOT, Stage 1 | 2 | 29 | 21
  Pubic Hair (Female): EOT, Stage 2: number analyzed (Participants) | 50 | 37 | 21
  Pubic Hair (Female): EOT, Stage 2 | 2 | 5 | 0
  Pubic Hair (Female): EOT, Stage 3: number analyzed (Participants) | 50 | 37 | 21
  Pubic Hair (Female): EOT, Stage 3 | 6 | 2 | 0
  Pubic Hair (Female): EOT, Stage 4: number analyzed (Participants) | 50 | 37 | 21
  Pubic Hair (Female): EOT, Stage 4 | 10 | 1 | 0
  Pubic Hair (Female): EOT, Stage 5: number analyzed (Participants) | 50 | 37 | 21
  Pubic Hair (Female): EOT, Stage 5 | 30 | 0 | 0
  Pubic Hair (Female): FU-12, Stage 1: number analyzed (Participants) | 51 | 35 | 21
  Pubic Hair (Female): FU-12, Stage 1 | 2 | 24 | 21
  Pubic Hair (Female): FU-12, Stage 2: number analyzed (Participants) | 51 | 35 | 21
  Pubic Hair (Female): FU-12, Stage 2 | 1 | 7 | 0
  Pubic Hair (Female): FU-12, Stage 3: number analyzed (Participants) | 51 | 35 | 21
  Pubic Hair (Female): FU-12, Stage 3 | 8 | 3 | 0
  Pubic Hair (Female): FU-12, Stage 4: number analyzed (Participants) | 51 | 35 | 21
  Pubic Hair (Female): FU-12, Stage 4 | 8 | 1 | 0
  Pubic Hair (Female): FU-12, Stage 5: number analyzed (Participants) | 51 | 35 | 21
  Pubic Hair (Female): FU-12, Stage 5 | 32 | 0 | 0
  Pubic Hair (Female): FU-24, Stage 1: number analyzed (Participants) | 50 | 35 | 21
  Pubic Hair (Female): FU-24, Stage 1 | 2 | 24 | 20
  Pubic Hair (Female): FU-24, Stage 2: number analyzed (Participants) | 50 | 35 | 21
  Pubic Hair (Female): FU-24, Stage 2 | 0 | 6 | 1
  Pubic Hair (Female): FU-24, Stage 3: number analyzed (Participants) | 50 | 35 | 21
  Pubic Hair (Female): FU-24, Stage 3 | 8 | 1 | 0
  Pubic Hair (Female): FU-24, Stage 4: number analyzed (Participants) | 50 | 35 | 21
  Pubic Hair (Female): FU-24, Stage 4 | 9 | 4 | 0
  Pubic Hair (Female): FU-24, Stage 5: number analyzed (Participants) | 50 | 35 | 21
  Pubic Hair (Female): FU-24, Stage 5 | 31 | 0 | 0
  Breasts (Female): Baseline, Stage 1: number analyzed (Participants) | 52 | 38 | 24
  Breasts (Female): Baseline, Stage 1 | 1 | 29 | 24
  Breasts (Female): Baseline, Stage 2: number analyzed (Participants) | 52 | 38 | 24
  Breasts (Female): Baseline, Stage 2 | 5 | 6 | 0
  Breasts (Female): Baseline, Stage 3: number analyzed (Participants) | 52 | 38 | 24
  Breasts (Female): Baseline, Stage 3 | 6 | 3 | 0
  Breasts (Female): Baseline, Stage 4: number analyzed (Participants) | 52 | 38 | 24
  Breasts (Female): Baseline, Stage 4 | 17 | 0 | 0
  Breasts (Female): Baseline, Stage 5: number analyzed (Participants) | 52 | 38 | 24
  Breasts (Female): Baseline, Stage 5 | 23 | 0 | 0
  Breasts (Female): EOT, Stage 1: number analyzed (Participants) | 50 | 37 | 21
  Breasts (Female): EOT, Stage 1 | 1 | 25 | 21
  Breasts (Female): EOT, Stage 2: number analyzed (Participants) | 50 | 37 | 21
  Breasts (Female): EOT, Stage 2 | 2 | 9 | 0
  Breasts (Female): EOT, Stage 3: number analyzed (Participants) | 50 | 37 | 21
  Breasts (Female): EOT, Stage 3 | 6 | 2 | 0
  Breasts (Female): EOT, Stage 4: number analyzed (Participants) | 50 | 37 | 21
  Breasts (Female): EOT, Stage 4 | 14 | 1 | 0
  Breasts (Female): EOT, Stage 5: number analyzed (Participants) | 50 | 37 | 21
  Breasts (Female): EOT, Stage 5 | 27 | 0 | 0
  Breasts (Female): FU-12, Stage 1: number analyzed (Participants) | 51 | 35 | 21
  Breasts (Female): FU-12, Stage 1 | 1 | 20 | 21
  Breasts (Female): FU-12, Stage 2: number analyzed (Participants) | 51 | 35 | 21
  Breasts (Female): FU-12, Stage 2 | 2 | 11 | 0
  Breasts (Female): FU-12, Stage 3: number analyzed (Participants) | 51 | 35 | 21
  Breasts (Female): FU-12, Stage 3 | 5 | 2 | 0
  Breasts (Female): FU-12, Stage 4: number analyzed (Participants) | 51 | 35 | 21
  Breasts (Female): FU-12, Stage 4 | 15 | 2 | 0
  Breasts (Female): FU-12, Stage 5: number analyzed (Participants) | 51 | 35 | 21
  Breasts (Female): FU-12, Stage 5 | 28 | 0 | 0
  Breasts (Female): FU-24, Stage 1: number analyzed (Participants) | 50 | 35 | 21
  Breasts (Female): FU-24, Stage 1 | 1 | 20 | 20
  Breasts (Female): FU-24, Stage 2: number analyzed (Participants) | 50 | 35 | 21
  Breasts (Female): FU-24, Stage 2 | 0 | 10 | 1
  Breasts (Female): FU-24, Stage 3: number analyzed (Participants) | 50 | 35 | 21
  Breasts (Female): FU-24, Stage 3 | 6 | 3 | 0
  Breasts (Female): FU-24, Stage 4: number analyzed (Participants) | 50 | 35 | 21
  Breasts (Female): FU-24, Stage 4 | 13 | 2 | 0
  Breasts (Female): FU-24, Stage 5: number analyzed (Participants) | 50 | 35 | 21
  Breasts (Female): FU-24, Stage 5 | 30 | 0 | 0

18. Secondary Outcome: Treatment Phase: Growth and Development as Measured by Parental Height
Description: Mid-parental height was calculated as the average of the biological father's and mother's heights. For boys, the sex-adjusted mid-parental height was calculated by adding 2.5 inches or 6.5 cm to the mean of the parents' heights. For girls, 2.5 inches or 6.5 cm was subtracted from the mean of the parents' heights.
Time Frame: Day 1
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 53 | 39 | 23
cm | 170.5 [162.0 to 176.7] | 170.0 [163.7 to 178.6] | 168.7 [163.0 to 174.1]

19. Secondary Outcome: Treatment Phase: Change From Baseline in Growth and Development as Measured by Bone Age
Description: Bone age was determined based on x-ray of the left wrist, hand, and fingers. Baseline value is the last available value on or prior to first dose date of study drug.
Time Frame: Baseline; FU-24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
Number analyzed (Participants) | 102 | 73 | 41
years
  Baseline: number analyzed (Participants) | 102 | 72 | 40
  Baseline | 15.5 [13.5 to 17.0] | 7.8 [6.8 to 9.0] | 4.8 [4.2 to 5.5]
  Change From Baseline at FU-24: number analyzed (Participants) | 92 | 68 | 35
  Change From Baseline at FU-24 | 0.6 [0.0 to 1.0] | 1.0 [0.0 to 1.2] | 0.5 [0.0 to 1.1]

20. Secondary Outcome: Treatment Phase: Swallowability of SOF/VEL as Assessed by the Participant's Ability to Swallow SOF/VEL Placebo Tablets at Baseline
Description: A SOF/VEL FDC swallowability assessment was performed using placebo tablets at baseline.
Time Frame: Baseline
Population: Participants in the Full Analysis Set with available data were analyzed. Swallowability assessment was performed in 12 to <18 years old and 6 to < 12 Years old only.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old
Number analyzed (Participants) | 102 | 73
Participants
  SOF/VEL 400/100mg Placebo Tablet, Able to Swallow: number analyzed (Participants) | 102 | 1
  SOF/VEL 400/100mg Placebo Tablet, Able to Swallow | 92 | 1
  SOF/VEL 400/100mg Placebo, Not Able to Swallow: number analyzed (Participants) | 102 | 1
  SOF/VEL 400/100mg Placebo, Not Able to Swallow | 10 | 0
  SOF/VEL 200/50mg Placebo, Able to Swallow: number analyzed (Participants) | 10 | 73
  SOF/VEL 200/50mg Placebo, Able to Swallow | 10 | 72
  SOF/VEL 200/50mg Placebo, Not Able to Swallow: number analyzed (Participants) | 10 | 73
  SOF/VEL 200/50mg Placebo, Not Able to Swallow | 0 | 1

21. Secondary Outcome: Treatment Phase: Number of Participants With Acceptability of SOF/VEL as Measured by a Questionnaire to Assess Acceptability, Including Palatability at Day 1
Description: Acceptability was assessed by numeric response marked on line between numbers 0 - 100. Higher scores indicate better acceptability and/or palatability.
Time Frame: Day 1
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- 12 to <18 Years Old: Treatment Phase: 2 * SOF/VEL 200/50 mg (adult and smaller size tablets based on swallowability assessment) once daily for 12 weeks.
- 6 to < 12 Years Old: Treatment Phase: SOF/VEL FDC 200/50 mg tablets once daily for 12 weeks.
- 6 to <12 Years Old: Treatment Phase: SOF/VEL FDC 200/50 mg oral granules once daily for 12 weeks.
- 3 to < 6 Years Old: Treatment Phase: SOF/VEL FDC 200/50 mg oral granules once daily for 12 weeks for participants who weighed ≥ 17 kg.
- 3 to <6 Years Old: SOF/VEL FDC 150/37.5 mg oral granules once daily for 12 weeks for participants who weighed < 17 kg.
Arm/Group | 12 to < 18 Years Old | 12 to <18 Years Old | 6 to < 12 Years Old | 6 to <12 Years Old | 3 to < 6 Years Old | 3 to <6 Years Old
Number analyzed (Participants) | 91 | 11 | 72 | 1 | 29 | 12
Participants
  Taste, Participants Who Did Not Taste Study Drug: number analyzed (Participants) | 91 | 11 | 71 | 1 | 27 | 12
  Taste, Participants Who Did Not Taste Study Drug | 61 | 5 | 42 | 0 | 8 | 5
  Taste, Participants Who Marked > 60 to 100: number analyzed (Participants) | 91 | 11 | 71 | 1 | 27 | 12
  Taste, Participants Who Marked > 60 to 100 | 16 | 3 | 11 | 0 | 6 | 3
  Taste, Participants Who Marked 40 to 60: number analyzed (Participants) | 91 | 11 | 71 | 1 | 27 | 12
  Taste, Participants Who Marked 40 to 60 | 11 | 1 | 6 | 0 | 4 | 1
  Taste, Participants Who Marked 0 to < 40: number analyzed (Participants) | 91 | 11 | 71 | 1 | 27 | 12
  Taste, Participants Who Marked 0 to < 40 | 3 | 2 | 12 | 1 | 9 | 3
  Easy to Take, Participants Who Marked > 60 to 100: number analyzed (Participants) | 89 | 11 | 71 | 1 | 27 | 12
  Easy to Take, Participants Who Marked > 60 to 100 | 82 | 9 | 60 | 0 | 13 | 4
  Easy to Take, Participants Who Marked 40 to 60: number analyzed (Participants) | 89 | 11 | 71 | 1 | 27 | 12
  Easy to Take, Participants Who Marked 40 to 60 | 5 | 1 | 3 | 0 | 4 | 2
  Easy to Take, Participants Who Marked 0 to < 40: number analyzed (Participants) | 89 | 11 | 71 | 1 | 27 | 12
  Easy to Take, Participants Who Marked 0 to < 40 | 2 | 1 | 8 | 1 | 10 | 6

22. Secondary Outcome: Treatment Phase: Number of Participants With Acceptability of SOF/VEL as Measured by a Questionnaire to Assess Acceptability, Including Palatability at Week 12
Description: as for outcome 21
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 to < 18 Years Old | 12 to <18 Years Old | 6 to < 12 Years Old | 6 to <12 Years Old | 3 to < 6 Years Old | 3 to <6 Years Old
Number analyzed (Participants) | 91 | 11 | 72 | 1 | 29 | 12
Participants
  Taste, Participants Who Did Not Taste Study Drug: number analyzed (Participants) | 90 | 11 | 70 | 1 | 23 | 8
  Taste, Participants Who Did Not Taste Study Drug | 49 | 2 | 33 | 0 | 8 | 2
  Taste, Participants Who Marked > 60 to 100: number analyzed (Participants) | 90 | 11 | 70 | 1 | 23 | 8
  Taste, Participants Who Marked > 60 to 100 | 24 | 5 | 14 | 0 | 4 | 1
  Taste, Participants Who Marked 40 to 60: number analyzed (Participants) | 90 | 11 | 70 | 1 | 23 | 8
  Taste, Participants Who Marked 40 to 60 | 10 | 1 | 12 | 1 | 4 | 3
  Taste, Participants Who Marked 0 to < 40: number analyzed (Participants) | 90 | 11 | 70 | 1 | 23 | 8
  Taste, Participants Who Marked 0 to < 40 | 7 | 3 | 11 | 0 | 7 | 2
  Easy to Take, Participants Who Marked > 60 to 100: number analyzed (Participants) | 89 | 11 | 70 | 1 | 23 | 8
  Easy to Take, Participants Who Marked > 60 to 100 | 83 | 9 | 65 | 1 | 20 | 6
  Easy to Take, Participants Who Marked 40 to 60: number analyzed (Participants) | 89 | 11 | 70 | 1 | 23 | 8
  Easy to Take, Participants Who Marked 40 to 60 | 3 | 0 | 5 | 0 | 1 | 1
  Easy to Take, Participants Who Marked 0 to < 40: number analyzed (Participants) | 89 | 11 | 70 | 1 | 23 | 8
  Easy to Take, Participants Who Marked 0 to < 40 | 3 | 2 | 0 | 0 | 2 | 1
  Feel About Taking Pills, Who Marked > 60 to 100: number analyzed (Participants) | 88 | 11 | 70 | 1 | 23 | 12
  Feel About Taking Pills, Who Marked > 60 to 100 | 82 | 8 | 60 | NA — Data not applicable for the oral granules group. | NA — Data not applicable for the oral granules group. | NA — Data not applicable for the oral granules group.
  Feel About Taking Pills, Who Marked 40 to 60: number analyzed (Participants) | 88 | 11 | 70 | 1 | 23 | 12
  Feel About Taking Pills, Who Marked 40 to 60 | 3 | 1 | 7 | NA — Data not applicable for the oral granules group. | NA — Data not applicable for the oral granules group. | NA — Data not applicable for the oral granules group.
  Feel About Taking Pills, Who Marked 0 to < 40: number analyzed (Participants) | 88 | 11 | 70 | 1 | 23 | 12
  Feel About Taking Pills, Who Marked 0 to < 40 | 3 | 2 | 3 | NA — Data not applicable for the oral granules group. | NA — Data not applicable for the oral granules group. | NA — Data not applicable for the oral granules group.

ADVERSE EVENTS:
Time Frame: Adverse Events: From first dose through last dose of the study drug (Up to 12 weeks) plus 30 days; All-Cause Mortality: First dose date up to Posttreatment Week 24
Description: The Safety Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug (SOF/VEL FDC).
Arm/Group | 12 to < 18 Years Old | 6 to < 12 Years Old | 3 to < 6 Years Old
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/73 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/102 | 2/73 | 0/41
Other Adverse Events (participants affected / at risk) | 65/102 | 53/73 | 26/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 12 to < 18 Years Old (N=102) | 6 to < 12 Years Old (N=73) | 3 to < 6 Years Old (N=41)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12 to < 18 Years Old (N=102) | 6 to < 12 Years Old (N=73) | 3 to < 6 Years Old (N=41)
Abdominal pain (Gastrointestinal disorders) | 6 | 9 | 2
Abdominal pain upper (Gastrointestinal disorders) | 10 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 5
Nausea (Gastrointestinal disorders) | 17 | 5 | 0
Vomiting (Gastrointestinal disorders) | 9 | 12 | 11
Fatigue (General disorders) | 22 | 9 | 5
Pyrexia (General disorders) | 10 | 8 | 6
Nasopharyngitis (Infections and infestations) | 6 | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 7 | 2
Product use issue (Injury, poisoning and procedural complications) | 0 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Dizziness (Nervous system disorders) | 9 | 2 | 1
Headache (Nervous system disorders) | 30 | 11 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years.

DOCUMENTS (2):
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT03022981/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03022981/SAP_001.pdf